CLINICAL TRIAL: NCT06849453
Title: Effects of Exercise Snacks and Sprint Interval Training on Cardiovascular Function in Overweight Adults: A Randomized Controlled Trial
Brief Title: Effects of Exercise Snacks and Sprint Interval Training in Overweight Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EESSITOA
Record Dates: First submitted 2025-02-04; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Cardiovascular Function; Cardiorespiratory Fitness
Keywords: Exercise Snacks; Sprint Interval Training; Overweight Adults; Cardiovascular Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of exercise interventions, it is difficult to blind study caregivers and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exercise snacks group (Active Comparator)
  Interventions: Behavioral: Exercise snacks group
- Sprint interval training group (Active Comparator)
  Interventions: Behavioral: Sprint interval training group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Exercise snacks group — Exercise snacks on the stairs for 8 weeks.
  Arms: Exercise snacks group
Behavioral: Sprint interval training group — Sprint interval training on the stairs for 8 weeks.
  Arms: Sprint interval training group

SUMMARY:
Exploring the efficacy and acceptability of exercise snacks (ES) and sprint interval training (SIT) could provide time-efficient, low-barrier alternatives for individuals, especially those who, due to 'lack of time, environment, and equipment,' struggle to meet traditional physical activity recommendations. This research aims to investigate the effects of ES and SIT, of equal exercise volume, on overweight adults.

DETAILED DESCRIPTION:
Engaging in regular physical activity has been shown to induce a range of beneficial physiological and psychological adaptations, including improved cardiorespiratory fitness, body composition, cardiovascular function, and reductions in negative emotions. However, global participation rates in physical activity remain suboptimal, with little significant improvement. Interviews and surveys have identified several potential barriers to low physical activity levels, with limitations such as 'lack of time, equipment, and facilities' often cited as the main perceived obstacles. Therefore, exploring the minimum effective dose of exercise in real-world settings is essential.

This study will employ a randomized clinical trial to examine the effectiveness and acceptability of two low-volume, high-intensity stair climbing exercises in overweight adults. It adopts a single-blind, parallel randomized design, with the intervention commencing immediately after the initial evaluation and randomization, following a pre-treatment/post-test framework. Eligible participants were recruited via convenience sampling and randomly assigned to one of three groups (one control group and two experimental groups):

1. A control group that will not receive any treatment.
2. Two experimental groups (ES and SIT), which will undergo a stair climbing-based physical training program following the initial evaluation. The two exercise interventions are designed with equal exercise volume, with the only difference being the rest (recovery) time between stair sprints. All exercise sessions are conducted under the supervision of professionals.

The aim of this study is twofold: First, to explore the impact of ES and SIT on cardiorespiratory fitness, body composition, and cardiovascular function in overweight adults. Second, to examine the acceptability of two low-volume, high-intensity stair climbing exercises by assessing participants' (1) acceptability, (2) reactions during the interventions, (3) enjoyment and affective valence during exercise, and (4) intentions at the end.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 35 years;
* Overweight but not obese (BMI ≥24 and ≤ 28 kg/m2);
* Physically inactive (3 or less bouts of purposeful exercise per week);
* Ability to understand the research details and voluntarily sign the informed consent form;
* Non-smoker (for >5 years);
* Body weight has been stable over the past six months, with no recent weight gain or loss behaviors;
* Healthy (see exclusion criteria).

Exclusion Criteria:

* Any chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, peripheral arterial disease, insulin- or non-insulin dependent diabetes or other metabolic disorders - all ascertained through preliminary screening;
* Individuals with a history of bone, joint or neuromuscular problems or a current musculoskeletal injury ascertained through preliminary screening;
* Abnormal electrocardiogram (ECG) results;
* Currently taking medication that may affect physiological testing;
* Contraindications to exercise.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-02-24 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness | 8 weeks
  The change of maximal oxygen uptake (VO2max) before and after intervention.

SECONDARY OUTCOMES:
Body composition | 8 weeks
  The change of body composition indexes (including fat mas, lean body mass, percentage of body fat) before and after intervention.
Lipid profile | 8 weeks
  The changes in concentrations of high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, total cholesterol, and triglyceride before and after intervention.
Endothelial function | 8 weeks
  The change of brachial Flow-Mediated Dilation (FMD) before and after intervention. Endothelial function will be assessed by FMD.
Arterial stiffness | 8 weeks
  The changes of brachial-ankle pulse wave velocity and ankle brachial index before and after intervention.
Resting blood pressure | 8 weeks
  The change of blood pressure (including systolic and diastolic blood pressure) before and after intervention.
Resting heart rate | 8 weeks
  The change of resting heart rate before and after intervention.
Waist Circumference | 8 weeks
  The change of waist circumference before and after intervention.
Hip Circumference | 8 weeks
  The change of hip circumference before and after intervention.
Body Mass Index (BMI ) | 8 weeks
  The change of BMI before and after intervention. BMI is calculated from the formula, Weight (kg) / Height2 (m2).

OTHER OUTCOMES:
Acceptability of the intervention | 8 weeks
  Intervention acceptability will be assessed using a theoretical framework of acceptability (TFA) questionnaire, completed only at the follow-up assessment. The seven domains of the TFA, along with overall acceptability, are measured using an 8-item questionnaire. The scale scores range from 0 to 5 with high scores indicating greater acceptability, and the total score representing the mean average of 7 individual domains of acceptability (each also rated 0-5).
Physical Activity Enjoyment Scale (PACES) | 8 weeks
  A modified version of the PACES will be used, the PACES scale was modified by removing 1 irrelevant item ('I was very/not at all absorbed in the activity'). The 17 items are scored on a 7-point Likert scale, resulting in an overall enjoyment score between 17 (not enjoyable), 68 (neutral), and 119 (enjoyable).
Intention Questionnaire | 8 weeks
  Intention questionnaire will be used after the 8 weeks intervention by a seven-point scale ranging from "Most likely never do this form of physical activity again (1)" to "Will likely do this three times per week every week (7)".
Exercise Enjoyment Scale | 4 weeks and 8 weeks
  Exercise enjoyment scale will be measured before, middle, and after intervention. The form will be presented to participants on a scale of 1 = 'not at all' to 7 = 'extremely,' and they will be asked, 'How much did you enjoy this exercise session?'
Feeling Scale | 4 weeks and 8 weeks
  Feeling scale will be measured before, middle, and after intervention. The one-item Feeling Scale will be used to measure general affective valence (i.e., pleasure and displeasure), participants will respond to the question 'How are you feeling right now?' (-5 = very bad to +5 = very good)
Rating of perceived exertion (RPE) | 4 weeks and 8 weeks
  Participants' RPE will be immediately assessed by Borg's Category-Ratio 10 scale after training sessions before, middle, and after intervention. The scale scores range from 0 to 10, with higher scores indicating greater perceived exertion.
Heart rate | 4 weeks and 8 weeks
  Mean and maximum heart rate of the intervention group will be monitored during each sprint.
Depression Anxiety Stress Scale-21 (DASS-21) | 8 weeks
  DASS-21 will be used before and after intervention. The scale has 21 questions, each question required participants to rate their experiences on a 4-point scale, where 0 indicated "did not apply to me at all", 1 indicated "applied to me to some degree or some of the time", 2 indicated "applied to me to a considerable degree or a good part of the time", and 3 indicated "applied to me very much or most of the time". The total scale scores range from 0 to 63, with higher scores indicating worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China

IPD SHARING:
Plan to Share IPD: No